CLINICAL TRIAL: NCT00004897
Title: PFL-Alpha Chemotherapy Followed by Surgery or FHX for Early Stage Esophageal Cancer - A Pilot Project
Brief Title: Combination Chemotherapy and Interferon Alfa Followed by Surgery and/or Radiation Therapy in Treating Patients With Stage I, Stage II, or Stage III Esophageal Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Institutional Review Board requested termination - all patients deceased and no new accrual.
Sponsor: Northwestern University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: NU 94I1; NU-94I1; NCI-G00-1679
Record Dates: First submitted 2000-03-07; First posted 2004-07-26 (Estimated); Last update posted 2012-06-12 (Estimated); Status verified 2012-06

CONDITIONS: Esophageal Cancer
Keywords: stage I esophageal cancer; stage II esophageal cancer; stage III esophageal cancer; squamous cell carcinoma of the esophagus; adenocarcinoma of the esophagus
MeSH Terms: conditions — Esophageal Neoplasms; Esophageal Squamous Cell Carcinoma; Adenocarcinoma Of Esophagus | interventions — Interferon-alpha; Cisplatin; Fluorouracil; Hydroxyurea; Leucovorin; Radiotherapy

INTERVENTIONS:
Biological: recombinant interferon alfa
Drug: cisplatin
Drug: fluorouracil
Drug: hydroxyurea
Drug: leucovorin calcium
Procedure: conventional surgery
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Interferon alfa may interfere with the growth of cancer cells. Radiation therapy uses high-energy x-rays to damage tumor cells. Combining more than one drug and combining chemotherapy with interferon alfa, surgery, and/or radiation therapy may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of combination chemotherapy and interferon alfa followed by surgery and/or radiation therapy in treating patients who have stage I, stage II, or stage III esophageal cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine response rates, duration of response, and performance status in patients with stage I-III esophageal cancer after treatment with cisplatin, fluorouracil, interferon alfa, and leucovorin calcium. II. Determine toxicities of this regimen in these patients. III. Determine relapse and survival rates in this patient population treated with this regimen. IV. Determine response rates, duration of response, performance status, and relapse and survival rates for inoperable candidates in this patient population treated with this regimen followed by radiotherapy. V. Determine the toxicities of this regimen followed by radiotherapy in these patients. VI. Evaluate recurrence following this treatment regimen in this patient population. VII. Compare roentgenographic and ultrasound responses to histopathologic responses with this regimen in this patient population. VIII. Evaluate the effects of this regimen and its relation to the ability to achieve negative surgical margins and evaluate the extent of multifocality, nodal disease, tumor size, and tumor grade. IX. Determine the incidence of perioperative complications following this regimen, including surgical as well as operative time, blood loss, perioperative transfusions, and length of hospital stay.

OUTLINE: Patients receive leucovorin calcium IV continuously on days 1-5.5, interferon alfa subcutaneously daily on days 1-6, cisplatin IV over 6 hours on day 1, and fluorouracil IV continuously on days 1-5. Treatment continues every 21 days for 3 courses in the absence of unacceptable toxicity. Approximately 4 weeks after chemotherapy, esophagectomy is performed in patients without evidence of locally advanced unresectable esophageal cancer or distant metastases. Patients determined to have residual disease following esophagectomy will be considered for radiotherapy. Patients not undergoing esophagectomy receive chemoradiotherapy 21-28 days after completion of initial chemotherapy. Patients receive oral hydroxyurea every 12 hours on days 0-5 and fluorouracil IV continuously on days 1-5. Patients undergo radiotherapy to esophagus daily on days 1-5. Treatment continues every 14 days for 7 courses in the absence of unacceptable toxicity. Patients are followed every 6 months for 2 years.

PROJECTED ACCRUAL: Approximately 15-45 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically or cytologically proven stage I-III squamous cell carcinoma or adenocarcinoma of the esophagus and gastro-esophageal junction Unidimensionally measurable disease

PATIENT CHARACTERISTICS: Age: Not specified Performance status: ECOG 0-2 Life expectancy: At least 270 days Hematopoietic: WBC greater than 3,000/mm3 Granulocyte count greater than 1,000/mm3 Platelet count greater than 100,000/mm3 Hepatic: Bilirubin, alkaline phosphatase, and SGOT no greater than 2 times upper limit of normal (ULN) Renal: Creatinine less than 2.0 mg/dL Creatinine clearance greater than 50 mL/min Cardiovascular: No serious cardiovascular disease that would preclude study Other: No prior or concurrent malignancy within past 5 years except nonmelanoma skin cancer No serious chronic medical illness that would preclude study No acute or chronic unresolved infection Not pregnant

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: No prior chemotherapy Endocrine therapy: Not specified Radiotherapy: No prior radiotherapy Surgery: Not specified

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1999-10; Primary Completion 2007-07 (Actual); Study Completion 2007-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Claudia Tellez, MD, Study Chair — Hematology-Oncology Associates of Illinois
Locations (1):
- Robert H. Lurie Comprehensive Cancer Center, Northwestern University, Chicago, Illinois, United States